CLINICAL TRIAL: NCT01711931
Title: Comparison of Everolimus- and Biolimus-Eluting Stents With Everolimus-Eluting Bioresorbable Vascular Scaffold Stents
Acronym: EVERBIOII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Stéphane Cook, Prof, Principal Investigator, University of Freiburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 043/12-CER-FR
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2014-05

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; bioresorbable vascular scaffold stents; everolimus; biolimus
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Everolimus-eluting bioresorbable vascular scaffold stents (Active Comparator)
  Interventions: Device: Implantation of everolimus-eluting bioresorbable vascular scaffold stent
- Everolimus-eluting stent (Active Comparator)
  Interventions: Device: Implantation of everolimus-eluting stents
- Biolimus-eluting stent (Active Comparator)
  Interventions: Device: Implantation of biolimus-eluting stents

INTERVENTIONS:
Device: Implantation of everolimus-eluting bioresorbable vascular scaffold stent
  Arms: Everolimus-eluting bioresorbable vascular scaffold stents
Device: Implantation of everolimus-eluting stents
  Arms: Everolimus-eluting stent
Device: Implantation of biolimus-eluting stents
  Arms: Biolimus-eluting stent

SUMMARY:
The purpose of this study is to compare the efficacy and safety of everolimus- and biolimus-bluting stents with everolimus-eluting bioresorbable vascular scaffold stents.

The null hypothesis to be rejected is that there is no significant difference with regard to lumen late loss at 9 months and a clinical end point of death, myocardial infarction and TVR at 12 months between everolimus-eluting and biolimus-eluting stents and everolimus-eluting bioresorbable vascular scaffold stents.

ELIGIBILITY:
Inclusion Criteria:

* elective PCI
* ability and willingness to provide written informed consent

Exclusion Criteria:

* ST-elevation myocardial infarction in the previous 48 hours
* moderate to severe renal failure (defined as creatinine clearance of 30-60 ml/min and <30ml/min respectively)
* known or presumed hypersensitivity to heparin, antiplatelet drugs and hypersensitivity to contrast dye incontrollable with premedication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Lumen Late Loss | 9 months
  as assessed by quantitative coronary angiogram

SECONDARY OUTCOMES:
Device-oriented major adverse cardiac events | 6 months, 1, 2, 5 years
  The composite of cardiac death, myocardial infarction (not clearly attributable to a nontarget vessel) and target lesion revascularization
Patient-oriented major adverse cardiac events | 6 months, 1, 2, 5 years
  The composite of all-cause mortality, any myocardial infarction and any revascularization

OTHER OUTCOMES:
Stent thrombosis | up to 5 years
  possible, probable and definite stent thrombosis
Periprocedural Complications (occurring <48 hours after the Intervention) | Periprocedural
  Type 4A MI Dissection Perforation

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Cook, Professor, Study Chair — University of Freiburg; Mario Togni, Professor, Study Director — University of Freiburg; Serban Puricel, MD, Principal Investigator — University of Freiburg
Locations (1):
- Fribourg Cantonal Hospital, Fribourg, Switzerland

REFERENCES:
- [Result] Arroyo D, Togni M, Puricel S, Gerard B, Sonja L, Corpataux N, Villeneuve H, Boute E, Stauffer JC, Goy JJ, Cook S. Comparison of everolimus-eluting and biolimus-eluting coronary stents with everolimus-eluting bioresorbable scaffold: study protocol of the randomized controlled EVERBIO II trial. Trials. 2014 Jan 7;15:9. doi: 10.1186/1745-6215-15-9. PMID 24398143
- [Derived] Bengueddache S, Cook M, Lehmann S, Arroyo D, Togni M, Puricel S, Cook S. Ten-year clinical outcomes of everolimus- and biolimus-eluting coronary stents vs. everolimus-eluting bioresorbable vascular scaffolds-insights from the EVERBIO-2 trial. Front Cardiovasc Med. 2024 Sep 10;11:1426348. doi: 10.3389/fcvm.2024.1426348. eCollection 2024. PMID 39323753
- [Derived] Kallinikou Z, Arroyo D, Togni M, Lehman S, Corpataux N, Cook M, Muller O, Baeriswyl G, Stauffer JC, Goy JJ, Puricel SG, Cook S. Vascular response to everolimus- and biolimus-eluting coronary stents versus everolimus-eluting bioresorbable scaffolds--an optical coherence tomography substudy of the EVERBIO II trial. Swiss Med Wkly. 2016 Jan 14;146:w14274. doi: 10.4414/smw.2016.14274. eCollection 2016. PMID 26766027
- [Derived] Puricel S, Arroyo D, Corpataux N, Baeriswyl G, Lehmann S, Kallinikou Z, Muller O, Allard L, Stauffer JC, Togni M, Goy JJ, Cook S. Comparison of everolimus- and biolimus-eluting coronary stents with everolimus-eluting bioresorbable vascular scaffolds. J Am Coll Cardiol. 2015 Mar 3;65(8):791-801. doi: 10.1016/j.jacc.2014.12.017. PMID 25720622